CLINICAL TRIAL: NCT03520127
Title: A Multi-center Registry Study Evaluating Outcomes in Breast Biopsy With the Intact™ Breast Lesion Excision System (BLES)
Brief Title: A Registry Study Evaluating Outcomes in Breast Biopsy With the Intact™ Breast Lesion Excision System (BLES)
Status: Terminated | Type: Observational
Why Stopped: Product withdrawn from the market due to a shift in sponsor business focus
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: 63-10-2356
Record Dates: First submitted 2018-04-05; First posted 2018-05-09 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Breast Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females, 18 years of age or older: Females, 18 years of age or older, who will undergo the Intact procedure
  Interventions: Device: Intact Breast Lesion Excision System (BLES)

INTERVENTIONS:
Device: Intact Breast Lesion Excision System (BLES) — Intact BLES is an automated, percutaneous biopsy device capable of delivering a surgical quality specimen for histological review of breast abnormalities. It is uniquely suited to maintain lesion architecture within the biopsy sample, providing an opportunity for pathological assessment and the potential avoidance of an open surgical procedure.

SUMMARY:
The purpose of this registry study is to collect use and clinical outcomes data following breast lesion excision or sampling with the Intact BLES.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* BIRADS ≤ 5, as initially imaged
* Subject is willing and capable of providing informed consent and has a scheduled or planned breast lesion excision or sampling where the Intact BLES is expected to be used

Exclusion Criteria:

* Male
* Subjects with subglandular (pre-pectoral, or "single plane") breast implants
* Subjects with electronic implantable devices (such as pacemakers and defibrillators)
* Subjects who are contraindicated for surgery due to factors such as anti-coagulant use which cannot be safely reversed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone the Intact procedure that are female and 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Lesion BIRADS score | Weeks prior to the Intact procedure
  Diagnostic imaging result
Imaging lesion size | Weeks prior to the Intact procedure
  Measured in mm
Lesion histology | Weeks prior to the Intact procedure
  Lesion biopsy results
Tissue margin (as reported from histology) rate | Weeks after the Intact procedure, up to approximately 12 weeks
  Procedure margin vs. margin size, measured in mm
Underestimation rate | Weeks after the Intact procedure, up to approximately 12 weeks
  Compared to maximum lesion size, measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Sakakeeny, PhD, Study Director — Medtronic Surgical Technologies
Locations (7):
- United States (7):
  - Birmingham Breast Care, Birmingham, Alabama
  - Winship Cancer Institute-Emory St. Joseph's, Atlanta, Georgia
  - Dalton Surgical Group, Dalton, Georgia
  - Metro Surgical Associates Inc., Lithonia, Georgia
  - Holyoke Medical Center, Holyoke, Massachusetts
  - Nashville Breast Center, Nashville, Tennessee
  - The Breast Center at Chesapeake Regional Healthcare, Chesapeake, Virginia

IPD SHARING:
Plan to Share IPD: Undecided